CLINICAL TRIAL: NCT02282488
Title: Effect of the Level of Dietary Protein on the Infant Hormonal Profile and Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 05.14.INF
Record Dates: First submitted 2014-10-24; First posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Low protein formula (Experimental): Low protein formula
  Interventions: Other: Low protein formula
- Group 2: high protein formula (Experimental): High protein formula
  Interventions: Other: High protein formula
- Group Breastfeeding (No Intervention): Breastfeeding

INTERVENTIONS:
Other: Low protein formula
  Other Names: LoF
  Arms: Group 1: Low protein formula
Other: High protein formula
  Other Names: HiF
  Arms: Group 2: high protein formula

SUMMARY:
A double blind, controlled, randomized, single site clinical trial of 2 parallel groups (Low protein formula =LoF and High protein formula =HiF) with a breastfeeding group (BF) as reference from birth to 1 year of age and a follow up period from 1 year to 5 years of age.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to show that infants taking (from birth) either a formula with a low protein content (LoF) or breast milk will have an IGF-1 level, at 4 months, 25% lower to the IGF-1 measured in infants that received a high protein content formula (HiF).

The secondary objectives are: The hormonal profile; the Fat mass (FM) gain and the Lean mass (LM); the metabolomics and aminogramm during the first year of life.

Subjects are included in the study for a duration of 5 years. From birth to 4 months they are exclusively fed BF or FF. From 4 months of age they can start diversification, but they maintain the starter formulas until 12 months (the BF group will receive LoF). Subjects are then followed up until 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

. Healthy newborn infant

* Full term infant (= 37 weeks gestation; = 42 weeks gestation)
* Birth weight = 2500 g and < 4200 g
* Singleton birth
* Infant is = 7 days of age at the time of enrollment
* For the BF group: The infant's mother has elected to exclusively breastfeed her baby, from enrollment to 4 months of age For the FF groups: The infant's mother has elected to exclusively formula feed her baby, from enrollment to 4 months of age
* Having obtained his/her or his/her legal representative's consent

Exclusion Criteria:

* Newborn whose mother's BMI was normal (<20 or = 25) at start of pregnancy

  * Newborn whose mother had developed gestational diabetes during pregnancy
  * Newborn whose mother has diabetes of type-1 or type-2
  * Newborn whose mother smoked > 5 cigarettes / day during pregnancy
  * Newborn whose mother had a drug dependence during pregnancy
  * Newborn whose mother has a chronic infectious disease
  * Newborn whose parents / caregivers cannot be expected to comply with treatment
  * Newborn currently participating in another clinical trial

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2006-04; Primary Completion 2009-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Analysis of IGF-1 value | 4 months
  Analyse the IGF-1 value and compare it

SECONDARY OUTCOMES:
Hormonal profile analysis (Insulin, C-peptide, Glucose, octanoyl ghrelin, Leptin and IGF-1) | 2 weeks, 4 months and 12 months
  The following markers will be measured: Insulin, C-peptide, Glucose, octanoyl ghrelin, Leptin and IGF-1 (IGF-1 at 4 months constitutes the primary outcome of this trial).
DEXA scan as a measure of the body composition | 2 weeks, 4 months and 12 months
  Measure of the Fat Mass (FM) gain and at the variations in Lean Mass (LM) during the first year of age.
aminogramm analysis | 2 weeks, 4 months and 12 months
  amino acids analysis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Steenhout, MD, Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- Hôpital de la Croix-Rouse, Lyon, France

REFERENCES:
- [Derived] Gonzalez-Garay AG, Serralde-Zuniga AE, Medina Vera I, Velasco Hidalgo L, Alonso Ocana MV. Higher versus lower protein intake in formula-fed term infants. Cochrane Database Syst Rev. 2023 Nov 6;11(11):CD013758. doi: 10.1002/14651858.CD013758.pub2. PMID 37929831